CLINICAL TRIAL: NCT04850521
Title: Remote Monitoring of Interstitial Lung Disease to Provide Continuity of Care and Shielding From Risks Associated With In-clinic Assessment
Brief Title: Remote Monitoring of Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: patientMpower Ltd. (Industry)
Collaborators: Quiddity Health Ltd. (Unknown); Innovate UK (Other Government)
Responsible Party: Sponsor
Other Study IDs: ILD patientMpower 01
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Remote Patient Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Remote monitoring: Remote monitoring software + connected devices
  Interventions: Other: Remote monitoring

INTERVENTIONS:
Other: Remote monitoring — patient-facing app + connected spirometer + connected pulse oximeter + clinician view portal

SUMMARY:
As in-clinic pulmonary function testing is greatly restricted due to Coronavirus Disease 2019 (COVID19), alternative approaches to monitoring patients with long-term respiratory conditions need to be developed and assessed. This project will evaluate the feasibility of a remote monitoring programme designed for interstitial lung disease (ILD) [including idiopathic pulmonary fibrosis (IPF)] patients which includes patient-reported spirometry & pulse oximetry (to estimate lung airflow and oxygen levels in the blood).

Patients with a confirmed diagnosis of ILD will be asked to measure spirometry & pulse oximetry once/day for approximately three months. Each patient will be supplied with a spirometer & pulse oximeter for home use. There will be no other changes to patients' care. The clinical teams responsible for care of the patients will be able to view all patient-recorded data immediately after data are recorded by the patient. Feasibility of remote monitoring will be assessed by determining the proportion of patients who provide measurements at least 3 times/week and on at least 70% of days in the observation period. Patient engagement (Patient Activation Measure), changes in spirometry measurements over time and healthcare resource utilisation (e.g. number of in-clinic visits) will also be assessed. Other outcomes assessed will include estimation of the proportion of patients with significant decreases in lung function, number of occasions where critical alert values of physiological parameters are reported and number of interventions by healthcare professionals in response to observations or alerts from remote monitoring. Feedback from patients and healthcare providers on user experience will also be sought.

Learnings from this project will be used to assess the wider application of delivery of digitally-based remote monitoring in management of long-term respiratory conditions.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of interstitial lung disease
* Forced Vital Capacity ≥50% predicted (at most recent in-clinic spirometry test)
* owns a smartphone or tablet device
* has a mobile telephone number, email address and access to internet at home
* willing to allow home monitoring of their health including spirometry and pulse oximetry data
* understands how to use mobile technology (e.g. has downloaded and used other "apps" on their mobile device; uses email)
* demonstrates willingness to measure spirometry and pulse oximetry daily for the duration of the study
* fluent in English language
* Written informed consent.

Exclusion Criteria:

* serious concomitant conditions which place the patient at high risk of respiratory distress, making them unsuitable to be managed at home
* confusion which would limit the patient's understanding of the project or the measurement procedures
* current or recent (within last 6 weeks before baseline) participation in another clinical research project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of interstitial lung disease (including idiopathic pulmonary fibrosis)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Frequency of use ≥3 days/week | 90 days
  Proportion of patients recording measurements ≥3 days/week
Frequency of use on ≥70% of study days | 91 days
  Proportion of patients recording measurements on ≥70% of study days

SECONDARY OUTCOMES:
Health-related quality of life | 91 days
  EuroQol 5-dimension 5-level (EQ-E5-DL) health status
Patient engagement | 91 days
  Patient Activation Measure
Change in Forced Vital Capacity (FVC) | 91 days
  Proportion of patients with ≥10% decreased FVC vs. baseline
Frequency of patients with alert values of pulse oximetry oxygen saturation (SpO2) | 91 days
  Proportion of patients with pulse oximetry SpO2 <93% at any time
Frequency of alert values of pulse oximetry SpO2 per patient | 91 days
  Number of pulse oximetry SpO2 <93% values per patient
Adherence to study measurements | 91 days
  Number of days patients record spirometry/number of days in observation period
Frequency of use ≥1 day/week | 91 days
  Proportion of patients recording measurements ≥1 day/week
Frequency of use ≥5 days/week | 91 days
  Proportion of patients recording measurements ≥5 days/week

OTHER OUTCOMES:
Time reviewing remote data | 91 days
  Clinic time reviewing portal data/patient
Clinic/patient contacts | 91 days
  Number of clinic center contacts with patient
Clinic spirometry visits | 91 days
  Number of in-clinic spirometry visits
Hospital admissions | 91 days
  Number of hospital admissions

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - Imperial College NHS Healthcare Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Lancashire Teaching Hospitals NHS Foundation Trust, Preston

REFERENCES:
- [Derived] Barth S, Edwards C, Saini G, Haider Y, Williams NP, Storrar W, Jenkins G, Stewart I, Wickremasinghe M. Feasibility and acceptability of remotely monitoring spirometry and pulse oximetry as part of interstitial lung disease clinical care: a single arm observational study. Respir Res. 2024 Apr 15;25(1):162. doi: 10.1186/s12931-024-02787-1. PMID 38622608